CLINICAL TRIAL: NCT00104234
Title: A Multicenter, Multinational Open-Label Extension Study of Recombinant Human N-acetylgalactosamine 4-sulfatase (rhASB) in Patients With Mucopolysaccharidosis VI
Brief Title: Study of rhASB in Patients With Mucopolysaccharidosis VI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASB-03-06
Record Dates: First submitted 2005-02-24; First posted 2005-02-25 (Estimated); Results first posted 2009-03-06 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Mucopolysaccharidosis VI
MeSH Terms: conditions — Mucopolysaccharidosis VI | interventions — N-Acetylgalactosamine-4-Sulfatase

ARMS (2):
- rhASB/rhASB (Other): N-acetylgalactosamine 4-sulfatase
  Interventions: Drug: N-acetylgalactosamine 4-sulfatase
- Placebo/rhASB (Other)
  Interventions: Drug: Placebo/rhASB

INTERVENTIONS:
Drug: N-acetylgalactosamine 4-sulfatase
  Other Names: rhASB
  Arms: rhASB/rhASB
Drug: Placebo/rhASB
  Arms: Placebo/rhASB

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety of rhASB treatment in patients with Mucopolysaccharidosis VI.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Patient must have successfully completed study ASB-03-05, including having received at least 20 of 24 scheduled weekly infusions and having missed no more then two consecutive infusions
* If female of childbearing potential, patient must have a negative pregnancy test

Exclusion Criteria:

* Pregnant or lactating patient
* Patient has received an investigational drug within 30 days prior to study enrollment
* Patient is unwilling or unable to travel to the primary site for periodic assessments

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-02; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BioMarin Pharmaceutical Inc., Novato, California, United States

REFERENCES:
- [Derived] Tandon PK, Kakkis ED. The multi-domain responder index: a novel analysis tool to capture a broader assessment of clinical benefit in heterogeneous complex rare diseases. Orphanet J Rare Dis. 2021 Apr 19;16(1):183. doi: 10.1186/s13023-021-01805-5. PMID 33874971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Global study sites were hospitals and medical clinics.
  First Enrollment: 05FEB04
  Last Dose: 28SEP06
Groups:
- rhASB/rhASB: Patients received rhASB in the double-blind study(ASB-03-05, NCT00067470)and continued to receive rhASB in the extension study(ASB-03-06).
- Placebo/rhASB: Patients received placebo in the double-blind study (ASB-03-05, NCT00067470)then received rhASB in the extension study (ASB-03-06).
Period: Overall Study
Arm/Group | rhASB/rhASB | Placebo/rhASB
Started | 19 | 20
Completed | 19 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhASB/rhASB | Placebo/rhASB | Total
Number analyzed (Participants) | 19 | 20 | 39
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic and baseline characteristics were recorded at baseline in the double-blind study, ASB-03-05.
  years
    Age | 13.7 (6.47) | 10.7 (4.35) | 12.2 (5.62)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic and baseline characteristics were recorded at baseline in the double-blind study, ASB-03-05.
  Participants
    Female | 12 | 14 | 26
    Male | 7 | 6 | 13
Race/Ethnicity, Customized [Number; unit: participants] — Demographic and baseline characteristics were recorded at baseline in the double-blind study, ASB-03-05.
  participants
    White, non-Hispanic | 15 | 9 | 24
    Hispanic | 1 | 3 | 4
    Black | 1 | 2 | 3
    Asian | 1 | 1 | 2
    Indigenous | 1 | 1 | 2
    Other | 0 | 4 | 4
Region of Enrollment [Number; unit: participants] — Demographic and baseline characteristics were recorded at baseline in the double-blind study, ASB-03-05.
  participants
    United States | 2 | 4 | 6
    Germany | 4 | 4 | 8
    United Kingdom | 3 | 3 | 6
    Brazil | 4 | 4 | 8
    France | 2 | 3 | 5
    Portugal | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: 12-Minute Walk Test
Description: Mean change in meters walked in 12 minutes. Mean change is the mean difference between the 12-Minute Walk Test at 96 weeks and that measured before first ever treatment with rhASB. For the rhASB/rhASB group, mean change is calculated for Week 96 - Baseline. For the placebo/rhASB group, mean change is calculated for Week 96 - Week 24.
Time Frame: Baseline of ASB-03-05 through week 96 of ASB-03-06
Population: The efficacy analysis included all subjects who continued in the extension study (ASB-03-06) except the 1 subject from the rhASB/rhASB group and 1 subject from the placebo/rhASB group who missed the Week 96 measurement.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | rhASB/rhASB | Placebo/rhASB
Number analyzed (Participants) | 18 | 18
meters | 187 (187) | 118 (127)

2. Secondary Outcome: 3-Minute Stair Climb
Description: Mean change in number of stairs climbed per minute in 3 minutes. Mean change is the mean difference between the 3-Minute Stair Climb at 96 weeks and that measured before first ever treatment with rhASB. Mean change is calculated for Week 96 - Baseline for the rhASB/rhASB group and for Week 96 - Week 24 for the placebo/rhASB group.
Time Frame: Baseline ASB-03-05 through week 96 of ASB-03-06.
Population: The efficacy analysis included all subjects who continued in the extension study (ASB-03-06) except 1 subject from the placebo/rhASB group who missed the Week 96 measurement.
Measure: Mean (Standard Deviation); unit: stairs/min
Arm/Group | rhASB/rhASB | Placebo/rhASB
Number analyzed (Participants) | 19 | 18
stairs/min | 13.1 (16.1) | 11.1 (10.0)

3. Secondary Outcome: Change in Urinary Glycosaminoglycans (GAG) Level
Description: Mean change in urinary GAG level for the first 72 weeks of rhASB treatment. For the rhASB/rhASB group, mean change was calculated for Week 72 -Baseline. For the placebo/rhASB, mean change was calculated for Week 96 - Week 24.
Time Frame: 72 weeks
Population: rhASB/rhASB and placebo/rhASB groups were combined for the analysis, representing 72 weeks of rhASB treatment in each group.
Measure: Mean (Standard Deviation); unit: microgram/mg creatinine
Groups:
- All Participants (N=37): rhASB/rhASB and placebo/rhASB groups were combined for analysis.
Arm/Group | All Participants (N=37)
Number analyzed (Participants) | 37
microgram/mg creatinine | -231 (91)

ADVERSE EVENTS:
Groups:
- All Participants: rhASB/rhASB and placebo/rhASB groups were combined for analysis.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 14/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=38)
Body increased temperature (Investigations) | 1 (1)
Broncopneumopathy (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cardiac failure (Cardiac disorders) | 2 (2)
Cervical cord compression (Nervous system disorders) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1)
Corneal Abscess (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2)
Hip Dysplasia (Congenital, familial and genetic disorders) | 1 (1)
Hip surgery (Surgical and medical procedures) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia obstructive (Gastrointestinal disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Osteotomy (Surgical and medical procedures) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=38)
Ear infection (Infections and infestations) | 17 (17)
Nasopharyngitis (Infections and infestations) | 16 (16)
Upper respiratory tract infection (Infections and infestations) | 15 (15)
Gastroenteritis (Infections and infestations) | 12 (12)
Bronchitis (Infections and infestations) | 9 (9)
Otitis externa (Infections and infestations) | 8 (8)
Influenza (Infections and infestations) | 7 (7)
Otitis media acute (Infections and infestations) | 7 (7)
Sinusitis (Infections and infestations) | 6 (6)
Hordeolum (Infections and infestations) | 5 (5)
Pharyngitis (Infections and infestations) | 5 (5)
Laryngitis (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 4 (4)
Dental Caries (Infections and infestations) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3)
Tinea pedis (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 6 (6)
Varicella (Infections and infestations) | 3 (3)
Bronchopneumonia (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 2 (2)
Fungal infection (Infections and infestations) | 2 (2)
Furuncle (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (28)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pulmonary hypertention (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 21 (21)
Vomiting (Gastrointestinal disorders) | 18 (18)
Abdominal pain (Gastrointestinal disorders) | 15 (15)
Nausea (Gastrointestinal disorders) | 11 (11)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6)
Toothache (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 27 (27)
Dizziness (Nervous system disorders) | 5 (5)
Paraesthesia (Nervous system disorders) | 4 (4)
Hyperreflexia (Nervous system disorders) | 3 (3)
Hypoaesthenia (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 3 (3)
Cervical myelopathy (Nervous system disorders) | 2 (2)
Migrane (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Pyrexia (General disorders) | 24 (24)
Fatigue (General disorders) | 8 (8)
Influenza like illness (General disorders) | 8 (8)
Chest pain (General disorders) | 7 (7)
Pain (General disorders) | 4 (4)
Hernia pain (General disorders) | 3 (3)
Infusion site pain (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 3 (3)
Rigors (General disorders) | 3 (3)
Athralgia (Musculoskeletal and connective tissue disorders) | 19 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Hip deformity (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertibral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint contracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Rash papular (Skin and subcutaneous tissue disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Prurigo (Skin and subcutaneous tissue disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Exanthem (Skin and subcutaneous tissue disorders) | 2 (2)
Face oedema (Skin and subcutaneous tissue disorders) | 2 (2)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 7 (7)
Eye irritation (Eye disorders) | 4 (4)
Eye pain (Eye disorders) | 4 (4)
Eye redness (Eye disorders) | 4 (4)
Visual acuity reduced (Eye disorders) | 4 (4)
Eyelid oedema (Eye disorders) | 2 (2)
Glaucoma (Eye disorders) | 2 (2)
Keratoconjunctivitis sicca (Eye disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 13 (13)
Hypoacusis (Ear and labyrinth disorders) | 7 (7)
Otorrhoea (Ear and labyrinth disorders) | 7 (7)
Cerumen impaction (Ear and labyrinth disorders) | 3 (3)
Post procedural pain (Injury, poisoning and procedural complications) | 10 (10)
Head injury (Injury, poisoning and procedural complications) | 4 (4)
Procedural site reaction (Injury, poisoning and procedural complications) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Poor venous access (Vascular disorders) | 4 (4)
Haematoma (Vascular disorders) | 2 (2)
Hyperaemia (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Cardiac valve disease (Cardiac disorders) | 5 (5)
Atrial hypertrophy (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2)
Cyanosis (Cardiac disorders) | 2 (2)
Dilatation atrial (Cardiac disorders) | 2 (2)
Neutrophil count increased (Investigations) | 3 (3)
QRS axis abnormal (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Cardiac murmur (Investigations) | 2 (2)
Oxygen saturation decreased (Investigations) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2)
Abnormal behavior (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 3 (3)
Hepatomegaly (Hepatobiliary disorders) | 2 (2)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the results shall be made by Sponsor in a joint publication. If such a multicenter publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from their site individually, subject however to comply with the other terms of the agreement.